CLINICAL TRIAL: NCT02630511
Title: Asthma Exacerbations and Vascular Function
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alberta (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: Pro00047054
Record Dates: First submitted 2015-12-04; First posted 2015-12-15 (Estimated); Last update posted 2021-07-01 (Actual); Status verified 2021-06

CONDITIONS: Asthma
MeSH Terms: conditions — Asthma | interventions — Mannitol; Methacholine Chloride; RE1-silencing transcription factor; Exercise

STUDY DESIGN:
Intervention Model Description: Randomized double-blind cross over design
Who Masked: Participant, Outcomes Assessor

ARMS (2):
- Asthma Group (Experimental): Asthma group to receive mannitol, methacholine or placebo challenge tests
  Interventions: Drug: Mannitol; Drug: Methacholine; Drug: Placebo; Other: Rest; Other: Exercise
- Control Group (Experimental): Control group to receive mannitol, methacholine or placebo challenge tests
  Interventions: Drug: Mannitol; Drug: Methacholine; Drug: Placebo; Other: Rest; Other: Exercise

INTERVENTIONS:
Drug: Mannitol — Mannitol consists of inhaling 0 (empty capsule acting as a placebo), 5, 10, 20, 40, 80, 160, 160, and 160 mg mannitol, resulting in a maximum cumulative dose of 635 mg
  Other Names: Mannitol Challenge Test
Drug: Methacholine — Methacholine consists of inhaling 0.0625 mg/mL, 0.25 mg/mL, 1 mg/mL, 4 mg/mL, and 16 mg/mL
  Other Names: Methacholine Challenge Test
Drug: Placebo — Placebo consists of inhaling humidified air
  Other Names: Placebo Challenge Test
Other: Rest
Other: Exercise

SUMMARY:
Although asthma is a disease of the airways, research is now showing that asthmatics are more likely to develop cardiovascular disease (CVD) compared to non-asthmatics. Vascular dysfunction is seen in people at high risk of CVD and has been linked to inflammation. During an asthma attack, levels of inflammation in the whole body increase, which could potentially explain why asthmatics are at increased risk of CVD. By exercising, people can change the amount of inflammation in their bodies, improve vascular function, and thereby reduce the risk of CVD. In the proposed study the investigators will assess if asthma attacks lead to increased risk of CVD by evaluating inflammatory levels and vascular function before and after asthma attacks. The investigators will also evaluate if exercise reduces the cardiovascular risk following asthma attacks. The results from this study will help in understanding why asthmatics are at increased risk of CVD.

DETAILED DESCRIPTION:
BACKGROUND & SCOPE: While asthma is generally considered to be a disease of the airways, there are important systemic consequences which have predisposed people with asthma to become more likely to die from cardiovascular (CV) disease compared to non-asthmatics. Additional CV risks have been reported in people with severe asthma, and there is a relationship between reductions in lung function and cardiac death. To date, little is known in regards to the interaction between asthma exacerbations and CV risk.

Brachial flow-mediated dilation (FMD) is used as a non-invasive tool to evaluate endothelial function. Brachial FMD is impaired in people with coronary dysfunction, and has been shown to predict future CV events better than traditional CV risk factors. People with asthma have previously been shown to have impaired endothelial function compared to non-asthmatics, but the underlying mechanism(s) are unclear.

Chronic systemic inflammation is an established risk factor and predictor of future CV events, and levels of systemic inflammation has been shown to be increased in asthma and to be are related to disease severity. While systemic inflammation can directly impair vascular function, it is unknown how an asthma attack may affect vascular function and CV risk. Thus, to gain better understanding of the increased CV risks associated with asthma exacerbations, the first aim of this study is to evaluate how acutely increased pulmonary inflammation affects vascular function in people with asthma.

Physical inactivity has previously been associated with increased systemic inflammation, while higher levels of physical activity can reduce inflammation and vascular dysfunction. Acute exercise has been shown to modulate the systemic responses to inflammatory insults, and being more physically active is associated with better asthma symptoms but whether acute exercise influences the systemic responses to asthma exacerbations is unknown. The second aim is to assess the influence of acute exercise on the systemic and vascular responses to acute pulmonary inflammation in asthma.

OBJECTIVE 1: To examine the acute impact of pulmonary inflammation and bronchoconstriction on systemic inflammation and vascular function in asthma.

METHODS & PROCEDURES, objective 1: Outline: Asthmatics will undergo a screening and three trials for which they will report to the laboratory in the morning of two consecutive days (Day 1 and Day 2) per trial. The screening day is to establish presence/absence of asthma and and will consist of pulmonary function testing before and after inhalation of a bronchodilator (Salbutamol), and an exercise challenge and cardiopulmonary fitness test. On Day 1, baseline pulmonary function and vascular function will be evaluated, and venous blood samples and exhaled breath condensate will also be obtained for evaluation of baseline systemic and pulmonary inflammation, respectively. The participants will then undergo either a mannitol challenge (Trial 1), a methacholine challenge (Trial 2), or a placebo (saline) challenge (Trial 3). At 1 hour post-challenge, another set of vascular function measurements, and systemic and pulmonary inflammation measurements will be done. The participants will be asked to come back 24 hours after each trial (Day 2) for a follow-up evaluation of vascular function and systemic inflammation. The order of the trials will be randomized and they will be separated by 1 week to allow for washout between tests.

Pulmonary function: A standard pulmonary function test will be performed by all participants as per established clinical guidelines.

Pulmonary inflammation: Exhaled breath condensate will be collected using RTube™ and analyzed for levels of CRP and markers of oxidative stress.

Systemic inflammation: The analysis of serum CRP, IL-6, TNFα, and nitrates and nitrites levels will be outsourced to Eve Technologies, Calgary.

Vascular function: Flow-mediated dilation (FMD) of the brachial artery following 5 minutes of forearm occlusion will be measured ultrasound imaging using our ultrasound machine. FMD will be determined using Doppler ultrasound immediately after the release of the occlusion. The secondary outcome is arterial stiffness, which will be determined using carotid - femoral/brachial pulse wave velocity, and PWV will be calculated from measurements of pulse transit time and the distance traveled by the pulse between recording sites.

Mannitol, methacholine and placebo challenge: Mannitol challenges have been shown to induce pulmonary inflammation in addition to bronchoconstriction in asthmatics and will be performed until either a cumulative dose of 635 mg has been obtained or until there is a reduction in the forced expiratory volume in the first second (FEV1) of ≥10% of baseline values. If bronchoconstriction occurs, the FEV1 will be monitored every 10 minutes until spontaneous recovery to within 5% of baseline FEV1, or reversed using 4 puffs (100 mg/puff) Salbutamol. Peripheral oxygen saturation will be monitored throughout the test. A methacholine challenge causes bronchoconstriction without an increase in pulmonary inflammation in asthmatics and will be used to separate between the effects of bronchoconstriction and pulmonary inflammation on vascular function. Except for the inhalation of methacholine, which will be performed according to established guidelines (in incremental concentrations until either 16 mg/ml methacholine has been inhaled, or there is a 20% reduction in FEV1), the same protocol will be used for the methacholine challenge and the placebo challenges. The participants will be blinded to the order of the tests.

OBJECTIVE 2: To evaluate the influence of acute exercise on systemic inflammatory and vascular responses to acute pulmonary inflammation.

METHODS & PROCEDURES, objective 2: Outline: The design of Objective 2 will be similar to the Mannitol challenge day in Objective 1 except the participants will in random order either a) exercise and inhale mannitol, b) exercise and placebo (saline), c) rest and inhale mannitol, or d) rest and placebo (saline). In addition to the inflammatory markers measured in Objective 1, the anti-inflammatory cytokine IL-10 will be measured in serum at each time point (baseline, 1 hour post-challenge, and 1 day post-challenge).

The exercise work load on the challenge day will correspond to 25 watts below achieved workload at anaerobic threshold during the screening day cardiopulmonary fitness test and will be held for 30 minutes. For the inactive day, the participants will be asked to withhold any exercise and/or moderate to heavy physical activity for 48 hours prior to the test. On the resting trial day, the participant will report to the lab at the same time of day as for exercise and instead rest quietly during for the same duration as the exercise period.

ELIGIBILITY:
Inclusion Criteria:

* Asthmatics, defined according to ATS and GINA guidelines,
* BMI <35kg/m2
* No known cardiovascular disease
* ACQ score equal to or less than 1.5 (controlled or partly controlled asthma)
* People without asthma (controls) will be recruited from the general population according to the same criteria, but with no history of asthma.

Exclusion Criteria:

* Pregnancy

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 52 (Actual)
Dates: Start 2015-12 (Actual); Primary Completion 2020-12 (Actual); Study Completion 2020-12 (Actual)

PRIMARY OUTCOMES:
Change from baseline flow-mediated dilation (FMD) to 15 minutes and 1 hour following bronchial challenge | At baseline, 15 min, 1 hour, and 24 hours following each intervention
  Flow-mediated dilation (FMD) of the brachial artery following 5 minutes of forearm occlusion will be measured using ultrasound (8L-RS 4.0-13.0 MHz probe, Vivid q, GE Healthcare, Mississauga, ON) and FMD data will be analyzed using FDA approved software available from Medical Imaging Applications (Coralville, IA, USA). FMD will be calculated as: (peak hyperemic diameter-baseline diameter)/baseline diameter x 100. FMD will be normalized for baseline diameter. Peak hyperemic brachial arterial velocity (and subsequently shear stress) will be determined using Doppler ultrasound, and used for normalization of FMD.

SECONDARY OUTCOMES:
Change from baseline arterial stiffness (cPWV) to 15 minutes and 1 hour following bronchial challenge | At baseline, 15 min, 1 hour, and 24 hours following each intervention
  Arterial stiffness will be determined using carotid - femoral pulse wave velocity (cPWV), and PWV will be calculated from measurements of pulse transit time and the distance traveled by the pulse between recording sites.
Change from baseline arterial stiffness (pPWV) to 15 minutes and 1 hour following bronchial challenge | At baseline, 15 min, 1 hour, and 24 hours following each intervention
  Arterial stiffness will be determined using carotid - radial pulse wave velocity (pPWV), and PWV will be calculated from measurements of pulse transit time and the distance traveled by the pulse between recording sites.
Change from baseline systemic inflammation to 15 minutes and 1 hour following bronchial challenge | At baseline, 15 min, 1 hour, and 24 hours following each intervention
  Serum analysis of inflammatory markers (i.e. of IL-6, IL-8, TNFα, and CRP).
Change from baseline pulmonary inflammation to 15 minutes and 1 hour following bronchial challenge | At baseline, 15 min, 1 hour, and 24 hours following each intervention
  Exhaled breath condensate (EBC) will be collected for analysis of CRP and 8-isoprostane.

CONTACTS AND LOCATIONS:
Overall Officials: Michael K Stickland, PhD, Principal Investigator — University of Alberta
Locations (1):
- Clinical Physiology Research Laboratory, Edmonton, Alberta, Canada

REFERENCES:
- [Derived] Moore LE, Brotto AR, Fuhr DP, Rosychuk RJ, Wong E, Bhutani M, Stickland MK. Impact of airway challenges on cardiovascular risk in asthma - a randomized controlled trial. PLoS One. 2023 Jul 17;18(7):e0288623. doi: 10.1371/journal.pone.0288623. eCollection 2023. PMID 37459335